CLINICAL TRIAL: NCT03068546
Title: Long Term Stability of Oral Microbiome Samples
Brief Title: Long-Term Stability of Oral Microbiome Samples
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999917062; 17-C-N062
Record Dates: First submitted 2017-02-28; First posted 2017-03-03 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Oral Microbiota; Long Term Sample Stability
Keywords: Oral Microbiota

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Participants providing samples: NCI employees agreeing to provide samples for microbiome sample study

SUMMARY:
Background:

The human biome is the collection of microbial genes found in and on the body. It has been associated with many health conditions. But certain factors might affect the findings from microbiome studies. These include collection method, lab handling, and data processing. Researchers want to test the effect of long-term storage in a freezer on two oral sample collections methods. These methods are OMNIgene ORAL and Scope mouthwash.

Objective:

To test the effect of long-term freezing on the oral microbiome measured from OMNIgene ORAL and Scope mouthwash.

Eligibility:

Employees of the National Cancer Institute who:

* Are age 18 or older
* Have not used antibiotics in the past 3 months

Design:

Participants will have 6 visits within 2 weeks. At visit 1 they will complete a questionnaire about health and lifestyle. All visits last 15-30 minutes and include:

* 1-2 saliva samples using OMNIgene ORAL: They will spit in a collector.
* 1-2 Scope samples: They will gargle with Scope mouthwash and spit in a cup.
* Questions about how well they followed the preparation procedures

Participants will follow preparation procedures: For 12 hours before each visit, they must not:

* Brush their teeth
* Floss
* Use mouthwash
* Eat or drink anything other than water
* Chew gum
* Consume throat lozenges or candies
* Smoke or chew tobacco

Participants samples will be stored in a freezer. They will get data about their oral microbiome if they wish.

DETAILED DESCRIPTION:
The human microbiome (i.e., the collection of microbial genes found in and on the human body) has been observed to be associated with numerous health conditions, but current methodological studies suggest that collection method, laboratory handling, bioinformatic processing of the data, and other factors can greatly affect microbiome study findings. In cohort studies, samples are typically collected at baseline, but are often not processed until sufficient cases have accumulated. This type of study design will require that samples remain frozen for likely many years prior to laboratory handling for microbiome measurements. To our knowledge, no study has considered the impact of long term storage of oral samples on oral microbiome characteristics. Therefore, we will evaluate the effect of long term storage of two oral sample collection methods (OMNIgene ORAL and Scope mouthwash) from 30 individuals who work at the NCI on oral microbiome characteristics. We will request that each participant will provide samples on 6 separate days over the course of two weeks. Participants will also fill out a short questionnaire. We will create aliquots from the pooled OMNIgene ORAL and Scope mouthwash samples from each individual, and immediately extract the DNA one aliquot. The remaining aliquots will be frozen at -80 degrees C and DNA will be extracted after one month, three months, six months, and one year after collection. The remaining aliquots will remain in the -80 degress C freezer for even longer term testing and other future studies. We will compare the microbial profiles from the stored samples to the immediately extracted samples to determine the effect of storage on oral samples.

ELIGIBILITY:
* ELIGIBILITY:

Anyone working at the NCI is eligible.

Children (<18 years of age) will not be included since children do not work for NCI and followup would be more difficult.

People of any age (adult), race, gender, or other factor are invited to participate.

No competent adult volunteers will be excluded.

The only exclusion of adults will be if the participant has taken antibiotic medication in the prior 3 months since antibiotic use has been shown to disrupt the oral microbiome, although less so than the fecal microbiome.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Employees of National Cancer Institute
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-06-29 (Actual); Primary Completion 2019-01-22 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Oral microbiome characteristics | One month after recruitment
  Microbial community characteristics

SECONDARY OUTCOMES:
Stability of oral microbiome characteristics | One year after recruitment
  Stability of oral microbial community over time

CONTACTS AND LOCATIONS:
Overall Officials: Christian Abnet, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Carroll IM, Ringel-Kulka T, Siddle JP, Klaenhammer TR, Ringel Y. Characterization of the fecal microbiota using high-throughput sequencing reveals a stable microbial community during storage. PLoS One. 2012;7(10):e46953. doi: 10.1371/journal.pone.0046953. Epub 2012 Oct 5. PMID 23071673
- [Background] Vogtmann E, Goedert JJ. Epidemiologic studies of the human microbiome and cancer. Br J Cancer. 2016 Feb 2;114(3):237-42. doi: 10.1038/bjc.2015.465. Epub 2016 Jan 5. PMID 26730578
- [Background] Zaura E, Brandt BW, Teixeira de Mattos MJ, Buijs MJ, Caspers MP, Rashid MU, Weintraub A, Nord CE, Savell A, Hu Y, Coates AR, Hubank M, Spratt DA, Wilson M, Keijser BJ, Crielaard W. Same Exposure but Two Radically Different Responses to Antibiotics: Resilience of the Salivary Microbiome versus Long-Term Microbial Shifts in Feces. mBio. 2015 Nov 10;6(6):e01693-15. doi: 10.1128/mBio.01693-15. PMID 26556275